CLINICAL TRIAL: NCT02531880
Title: Investigation of Blood-Brain-Barrier Breakdown Using Manganese Magnetic Resonance Imaging in Drug-Resistant Epilepsy
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 150177; 15-N-0177
Record Dates: First submitted 2015-08-22; First posted 2015-08-25 (Estimated); Last update posted 2025-12-31 (Actual); Status verified 2025-05-02

CONDITIONS: Epilepsy
Keywords: MRI; Manganese Enhanced MRI; Seizure Disorder; Seizures; Epileptic Focus
MeSH Terms: conditions — Epilepsy; Seizures | interventions — N,N'-bis(pyridoxal-5-phosphate)ethylenediamine-N,N'-diacetic acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- 1 (Experimental): Patients will be given the study drug
  Interventions: Drug: Mangafodipir

INTERVENTIONS:
Drug: Mangafodipir — Patients will be imaged interictally with a gadolinium enhanced MRI session. The administration of mangafodipir will be done as an inpatient during long-term video EEG recording, to ensure administration in the peri-ictal period.

SUMMARY:
Background:

- The blood-brain barrier separates the brain from the rest of the body. Epilepsy is a neurological disease that causes seizures. It can affect this barrier. Researchers think a contrast agent called mangafodipir might be better able to show areas of the brain that epilepsy affects.

Objective:

- To see if mangafodipir is well tolerated and safe. To see if it can show, on an MRI, areas of the brain that epilepsy affects.

Eligibility:

* People ages 18-60 who:
* Have epilepsy not controlled by drugs
* Prior or concurrent enrollment in 18-N-0066 is required

Design:

* Participants will be screened with:
* Medical history
* Physical exam
* Blood and urine tests
* Participants will have up to 6 visits in 1-3 months. Those with epilepsy will have an inpatient stay lasting 2-10 days. Visits may include:
* Video-EEG monitoring for participants with epilepsy
* An IV catheter put in place: a needle guides a thin plastic tube into an arm vein.
* Getting mangafodipir through the IV.
* 5 MRI scans over a 10-day period: a magnetic field and radio waves take pictures of the brain. Participants lie on a table that slides into a metal cylinder. They are in the cylinder for 45-90 minutes, lying still for up to 10 minutes at a time. The scanner makes loud knocking sounds. Participants will get earplugs.
* A final MRI at least 2 weeks after receiving mangafodipir. Gadolinium is given through an IV catheter....

DETAILED DESCRIPTION:
Objective:

The primary goals of this pilot study are to (1) describe the safety profile of administration of mangafodipir in patients with epilepsy and (2) investigate the prevalence of blood-brain barrier disruption (BBBD) in patients with drug-resistant focal epilepsy using peri-ictal manganese enhanced magnetic resonance imaging (MEMRI) and interictal gadolinium dynamic contrast-enhanced MRI (DCE-MRI) and determine if these methods will allow for visualization of seizure foci. Secondary objectives are further exploration of MEMRI and DCE-MRI properties in patients with epilepsy.

Study population:

40 patients with drug-resistant epilepsy.

Design:

Screening of enrolled participants will include a medical history, physical exam, blood and urine laboratory testing. There are two arms of this study; patients may be enrolled in either arm or both. For one arm, patients will be imaged interictally with a gadolinium enhanced MRI session (DCE-MRI). For the other arm, patients will be imaged peri-ictally with manganese enhanced MRI (MEMRI) as an inpatient during long-term video EEG recording, to ensure administration in the peri-ictal period. Patients will receive a baseline MRI scan, IV mangafodipir injection and will then be serially scanned with non-contrast MRI scans.

Outcome measures:

The primary outcomes are (1) description of the safety profile of mangafodipir administration in patients with epilepsy, and (2) evaluation of the utility of MEMRI and/or DCE-MRI in identifying focal BBBD in the seizure onset zone identified by standard clinical, EEG, and imaging studies, and the homologous contralateral region.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 18-60.
* Able to give written informed consent directly.
* Drug resistant epilepsy participants will be defined as having clinically documented seizures with consistent EEG evidence as defined by the 1981 International Classification of Epileptic Seizures, refractory to standard anti-seizure treatment for at least one year prior to enrolling in this study and with an average of at least one seizure per month. This criterion will be established by preliminary screening NINDS Epilepsy Service under protocol 18-N-0066. Seizure focus localization will be determined by standard clinical, neurophysiologic, and imaging studies. Prior or concurrent enrollment in 18-N-0066 is required.

EXCLUSION CRITERIA:

General exclusions:

* Patients with epilepsy who are not surgical candidates
* Significant structural brain abnormality such as a brain tumor, stroke, brain damage from head trauma or blood vessel abnormalities, on the baseline MRI scan.
* Positive test for HIV
* Pregnancy or breast-feeding
* Claustrophobia to a degree that the subject would feel uncomfortable in the MRI machine.
* Cannot lie on their back for at least two hours.
* Risk for MRI scan, (e.g., any non-organic implant or other device such as a cardiac pacemaker or infusion pump or other metallic implants, objects or body piercings that cannot be removed, or history of being a welder or metal worker due to small metal fragments in the eye)
* Unwilling to allow sharing and/or use in future studies of coded data that are collected for this study

MEMRI component specific exclusions (applicable only to patients participating in this arm of the study):

* History of post-ictal psychosis or post-ictal aggression
* Planning to get pregnant in the next 2 months
* History of clinically significant liver or kidney disease that could potentially increase the risk of CNS damage due to manganese exposure
* A history of drug or alcohol abuse/dependence (subjects scoring 8 or higher on the AUDIT scale)
* Screening lab abnormalities demonstrating values more than 2 times the upper limit of normal for AST, ALT, bilirubin, alkaline phosphatase, BUN, creatinine
* Previous presumed occupational exposure to manganese (i.e., having worked in a mine, foundry, smelter, dry cell battery manufacturing facility, or agriculture)
* Allergy to manganese
* On-going treatment with calcium-channel blocker
* Iron-deficiency anemia
* Personal history of Parkinson s Disease or Parkinsonism or presence of this disease in a 1st degree relative

Gadolinium enhanced MRI component specific exclusions (applicable only to patients participating in this arm of the study):

* Estimated GFR <60, tested within 1 week of scan
* Allergy to gadolinium

Of note, patients who are ineligible for one arm of the study may still be eligible for and participate in the other arm of the study.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-11-19 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
evaluation of the utility of MEMRI and/or DCE-MRI in identifying focal BBBD in the seizure onset zone identified by standard clinical, EEG, and imaging studies, and the homologous contralateral region. | after mangafodipir administration
  evaluation of the utility of MEMRI and/or DCE-MRI in identifying focal BBBD in the seizure onset zone identified by standard clinical, EEG, and imaging studies, and the homologous contralateral region.
description of the safety profile of mangafodipir administration in patients with epilepsy | after mangafodipir adminstration
  safety profile

CONTACTS AND LOCATIONS:
Overall Officials: Sara K Inati, M.D., Principal Investigator — National Institute of Neurological Disorders and Stroke (NINDS)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2015-N-0177.html